CLINICAL TRIAL: NCT07043192
Title: The Role of Venous-to-Arterial PCO₂ Gap and Critical Closing Pressure in Fluid Resuscitation Evaluation and Hemodynamic Evaluation in Patients With Sepsis Shock
Brief Title: Critical Closing Pressure and PCO₂ Gap in Fluid Resuscitation for Septic Shock
Status: Active, not recruiting | Type: Observational
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Shitong Diao, Principal Investigator, Peking Union Medical College
Other Study IDs: K8248
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Septic Shock; Fluid Resuscitation; Tissue Perfusion Pressure; Carbon Dioxide Pressure
Keywords: septic shock; fluid resuscitation; tissue perfusion pressure; carbon dioxide pressure
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fluid responsiveness positive: The determination of an increase of ≥10% in cardiac output before and after expansion.
- fluid responsiveness negetive: The determination of an increase of <10% in cardiac output before and after expansion.

SUMMARY:
This study is based on the following key hypotheses:

PvaCO₂ (Venous-to-Arterial CO₂ Gap) Hypothesis:

Changes in PvaCO₂ (ΔPvaCO₂) following fluid resuscitation correlate with changes in cardiac output (CO) and can serve as a reliable predictor of fluid responsiveness in septic shock patients.

The relationship between PvaCO₂ and CO is influenced by metabolic factors (VCO₂), hemodynamic status, and the Haldane effect (oxygenation-dependent CO₂ binding to hemoglobin).

Pcrit (Critical Closing Pressure) & TPP (Tissue Perfusion Pressure) Hypothesis:

Elevated Pcrit and reduced TPP (TPP = MAP - Pcrit) are associated with impaired microcirculatory flow and worse clinical outcomes (e.g., 28-day mortality, organ dysfunction).

Restoring the "vascular waterfall" phenomenon (Pcrit > mean systemic filling pressure) may improve macrocirculation-microcirculation coupling and tissue oxygenation.

2. Study Design Overview 2.1 Study Type Prospective observational cohort with a retrospective validation arm using external databases (e.g., MIMIC-IV).

Single-center study (Peking Union Medical College Hospital ICU). 2.2 Study Population Inclusion Criteria Adults (18-80 years) with septic shock (Sepsis-3 criteria + vasopressor-dependent hypotension + lactate >2 mmol/L).

Requires invasive hemodynamic monitoring (arterial line, central venous catheter).

Undergoing fluid challenge (clinically indicated). Exclusion Criteria Pregnancy, non-septic shock (e.g., cardiogenic), mechanical circulatory support (ECMO/IABP).

Severe COPD, intracardiac shunts, or conditions interfering with CO₂/VO₂ measurements.

2.3 Interventions & Measurements Fluid Resuscitation Protocol 500 mL 4% gelatin infused over 15 min (pressure bag at 300 mmHg). Hemodynamic/metabolic data collected pre- and post-fluid challenge (within 10 min).

Key Data Collected

Hemodynamics:

MAP, CVP, CO (PiCCO/ultrasound), Pcrit (derived from MAP-CO curve fitting). TPP = MAP - Pcrit.

Metabolic Parameters:

PvaCO₂, CvaCO₂, VCO₂, VO₂ (Es-COVX module). Lactate, ScvO₂, Hb, arterial/venous blood gases.

Outcomes:

Primary: 28-day mortality. Secondary: Lactate clearance, AKI incidence, ICU length of stay, vasopressor requirements.

DETAILED DESCRIPTION:
1. Study Background Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection, with septic shock being a subset of sepsis. Septic shock is defined as persistent hypotension requiring vasopressors to maintain a mean arterial pressure (MAP) ≥65 mmHg and serum lactate >2 mmol/L despite adequate fluid resuscitation. The mortality rate associated with sepsis ranges from 13.1% to 35.5%, and its increasing incidence has led to significant healthcare resource utilization and economic burden. Early recognition and timely treatment are critical for patients with sepsis and septic shock.

   Hemodynamics play a central role in sepsis resuscitation. The core issue in shock is inadequate cellular oxygen utilization, making the goal of shock therapy to increase oxygen delivery to meet demand and address systemic hypoperfusion. Carbon dioxide (CO₂), as a byproduct of cellular oxygen metabolism, has garnered attention.

   The venous-to-arterial CO₂ gap (PvaCO₂) and critical closing pressure (Pcrit) are emerging as potential markers for evaluating fluid responsiveness and tissue perfusion. However, their clinical utility remains controversial due to conflicting results and the influence of factors such as hemoglobin, pH, and the Haldane effect. This study aims to explore the dynamic changes in PvaCO₂ and CvaCO₂ during fluid resuscitation and investigate the role of Pcrit and tissue perfusion pressure (TPP) in risk stratification and blood pressure management for septic shock patients.
2. Study Objectives To evaluate the predictive value of ΔPvaCO₂ (change in PvaCO₂) for fluid responsiveness in septic shock patients.

   To assess the contributions of VCO₂, the Haldane effect, and cardiac output (CO) to changes in PvaCO₂ and CvaCO₂ during fluid resuscitation.

   To investigate the role of Pcrit and TPP in risk stratification and their potential as additional targets for blood pressure management in sepsis.
3. Methods and Procedures Study Design: Prospective observational study in ICU patients with septic shock.

Participants:

Inclusion Criteria:

Age 18-80 years.

Diagnosis of septic shock per Sepsis-3 criteria.

Requirement for invasive hemodynamic monitoring (arterial and central venous catheters).

Clinical indication for fluid challenge (e.g., hypotension, signs of hypoperfusion).

Exclusion Criteria:

Pregnancy or lactation.

Other types of shock (e.g., cardiogenic, obstructive).

Mechanical circulatory support (e.g., ECMO, IABP).

Severe respiratory or cardiovascular contraindications.

Data Collection:

Demographics and Clinical Data: Age, gender, SOFA/APACHE II scores, infection source, comorbidities, 28-day mortality.

Laboratory Tests: Lactate, hemoglobin, ScvO₂, SaO₂, arterial/venous blood gases.

Hemodynamic Monitoring:

Continuous MAP, CVP, and CO measurements (via PiCCO or echocardiography).

VO₂ and VCO₂ monitoring using a metabolic cart.

Fluid Challenge: 500 mL of 4% gelatin administered over 15 minutes, with hemodynamic and metabolic measurements pre- and post-infusion.

Pcc and Pmsf Measurement Protocol :

Interrupt Spontaneous Breathing: Temporarily suspend patient-triggered ventilation to ensure controlled mechanical ventilation.Adjust Ventilator to Pressure Control (PC) Mode: Apply incremental airway pressures of 5, 15, 25, and 35 cmH₂O, each maintained for 12 seconds.

Hemodynamic Data Acquisition:

Continuous Cardiac Output (CCO): Recorded on a beat-to-beat basis and averaged over the 12-second interval (displayed on monitor).

Additional Parameters: Simultaneously measure:Arterial pressure (systolic, diastolic), Heart rate (HR), Central venous pressure (CVP),Repetition: Each pressure level is tested 3 times to ensure reproducibility.

Data Analysis:

CO-MAP Regression: Plot cardiac output (CO) against mean arterial pressure (MAP) for each airway pressure.Pcrit Determination: The y-intercept of the CO-MAP curve represents critical closing pressure (Pcrit).CO-CVP Regression: Plot CO against CVP to derive mean systemic filling pressure (Pmsf) as the y-intercept.Pcrit and TPP: Derived from MAP-CO regression curves (TPP = MAP - Pcrit).

Measurement of VO₂ and VCO₂ Using Dräger Ventilators：1. Equipment Setup Ventilator Model: Dräger Evita V800, XLUNGE module (or equivalent with metabolic monitoring capabilities).

Required Accessories:

D-lite™ or Pediatric Flow Sensor: Installed between the endotracheal tube and ventilator circuit.

Gas Sampling Line: Connected to the flow sensor and ventilator's gas analyzer. Calibration Syringe: For flow sensor calibration. 2. Pre-Measurement Checks Calibration:Perform auto-calibration of the flow sensor and gas analyzer (follow ventilator prompts).

Verify O₂ and CO₂ sensor accuracy with known gas mixtures if available.

Circuit Integrity:

Ensure no air leaks around the endotracheal tube or sensor. Confirm gas sampling line is patent and dry (replace if contaminated with secretions).

3. Measurement Protocol

Stabilization Phase:

Maintain steady-state ventilation for ≥5 minutes (fixed FiO₂, PEEP, and tidal volume).

Pause endotracheal suctioning and discontinue humidification temporarily (water vapor interferes with gas analysis).

Data Acquisition:

Activate the XLUNGE metabolic module or equivalent. Select "Metabolic Monitoring" mode to display real-time VO₂ (O₂ consumption) and VCO₂ (CO₂ production).

Measurement Duration: Record values over ≥3 minutes to average respiratory cycle variability.

Key Parameters:

VO₂ (mL/min): Derived from O₂ uptake ([FiO₂ × inspired volume] - [FeO₂ × expired volume]).

VCO₂ (mL/min): Calculated from CO₂ elimination ([FeCO₂ × expired volume] - [FiCO₂ × inspired volume]).

Respiratory Quotient (RQ): Auto-calculated as VCO₂/VO₂.

Statistical Analysis:

Sample size: 48 patients (accounting for 20% dropout). Correlation analysis (Pearson/Spearman), ROC curves for predictive performance, and Cox regression for prognostic modeling.

4. Outcome Measures Primary Outcome: Change in cardiac output (CO) after fluid resuscitation. Secondary Outcomes: Lactate clearance, ICU length of stay, vasopressor requirements, 24-hour fluid balance.

5. Quality Control Standardized protocols for data collection and monitoring. Two independent physicians for eligibility assessment. Electronic medical record verification for baseline data.

6. Ethical Considerations Informed consent will be obtained from all participants or their legal representatives.

Patient data will be anonymized to ensure confidentiality.

The study complies with the Declaration of Helsinki and local regulatory requirements.

7. Statistical Methods Software: SPSS 27.0, GraphPad Prism 10.0, PASS 2021.

Tests: Shapiro-Wilk for normality, t-tests/Wilcoxon for group comparisons, ROC analysis for predictive accuracy.

Significance Level: P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.

Diagnosis of septic shock per Sepsis-3 criteria.

Requirement for invasive hemodynamic monitoring (arterial and central venous catheters).

Clinical indication for fluid challenge (e.g., hypotension, signs of hypoperfusion).

Exclusion Criteria:

* Pregnancy or lactation.

Other types of shock (e.g., cardiogenic, obstructive).

Mechanical circulatory support (e.g., ECMO, IABP).

Severe respiratory or cardiovascular contraindications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic shock patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | From enrollment to the end of treatment at 2 days
  Change in cardiac output (CO) after fluid resuscitation

SECONDARY OUTCOMES:
Lactate clearance | From enrollment to the end of treatment at 1 weeks
  The percentage decrease in lactic acid from the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China